CLINICAL TRIAL: NCT06392867
Title: Intermittent Theta-burst Stimulation for Major Depression: an Intensity-response Study
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: The Hong Kong Polytechnic University (Other)
Collaborators: Health and Medical Research Fund (Other Government)
Responsible Party: Principal Investigator, Dr Georg Kranz, Assistant Professor, The Hong Kong Polytechnic University
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Basic Science
Other Study IDs: HSEARS20221101008
Record Dates: First submitted 2024-04-23; First posted 2024-05-01 (Actual); Last update posted 2025-03-14 (Actual); Status verified 2025-03

CONDITIONS: Depression, Unipolar
Keywords: Transcranial magnetic stimulation, TMS; Major Depressive Disorder; iTBS; TMS treatment for depression
MeSH Terms: conditions — Depressive Disorder; Depressive Disorder, Major

STUDY DESIGN:
Intervention Model Description: Patients with Major Depressive Disorder will undergo daily intermittent theta-burst stimulation (iTBS) at left DLPFC, 20 sessions in 4 weeks. It is to investigate the potential antidepressant effects of iTBS treatment at a much lower stimulation intensity than the one currently employed by most centers in the United States and approved in these centers.
  The current study proposes a randomized, triple-arm, controlled trial to compare the efficacy of iTBS at 75% (iTBS75) and 120% (iTBS120) rMT with sham iTBS (SiTBS). Based on the following considerations, SiTBS was selected to be compared with iTBS75 and iTBS120: SiTBS will reveal placebo antidepressant effects and serve as a control.
Who Masked: Participant, Care Provider, Outcomes Assessor
Masking Description: Prior to the treatment, each participant will visit The Hong Kong Polytechnic University on a separate day. During the first visit, the researcher will also measure each participant's rMT. The PI will randomly assign the participant to different groups, such as sham group, 75% group, and 120% group, and calculate the maximum intensity of treatment based on the respective groups of the participant. To provide individualized treatment intensity to each participant, the TMS operator will receive the information from the PI and perform the treatment according to the determined intensity. The operator does not know the participant's rMT and sham coil is used. Furthermore, the participants have never received TMS treatment before taking part in this study, so they do not understand the difference between a placebo and a real treatment.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- SiTBS (Sham Comparator): The participants will not receive any benefit from the intermittent theta-burst stimulation (iTBS) if they use the inactive side of the coil.
  Interventions: Device: intermittent theta-burst stimulation (iTBS)
- iTBS75 (Active Comparator): The intensity of intermittent theta-burst stimulation (iTBS) applied to the participant will be 75% of their individual rest motor threshold (rMT).
  Interventions: Device: intermittent theta-burst stimulation (iTBS)
- iTBS120 (Active Comparator): The intensity of intermittent theta-burst stimulation (iTBS) applied to the participant will be 120% of their individual rest motor threshold (rMT).
  Interventions: Device: intermittent theta-burst stimulation (iTBS)

INTERVENTIONS:
Device: intermittent theta-burst stimulation (iTBS) — iTBS treatment will be performed as comprising 3-pulse 50-Hz bursts, applied every 200 ms (at 5 Hz). iTBS consists of 2-second trains with an inter-train-interval of 8 seconds. Repeat trains (30 pulses; 10 bursts) 20 times to reach a total number of 600 pulses (3x10x20) which equals the standard number of pulses in a daily iTBS treatment session, as approved by the FDA. The stimulation site over the left DLPFC will be determined using the international 10-20 system for EEG electrodes corresponding to the F3 location. 20 daily treatment sessions will be performed from Mondays to Fridays for four weeks for all included patients.
  Treatments will be performed at the brain stimulation laboratory at the Hong Kong Polytechnic University. Stimulation will be delivered using a MagPro X100 model (details about MagPro X100: magventure.com/en_eur/products/magpro-x100/ ) and a Cool-B65 A/P Butterfly Coil is used in this study.

SUMMARY:
The United States Food and Drug Administration (FDA) approved intermittent theta-burst stimulation (iTBS) in 2018 as a form of repetitive transcranial magnetic stimulation (rTMS). Hospitals worldwide use it to treat major depressive disorder (MDD). It is safe, effective, even for depressed patients unable to respond to standard pharmacological treatment and is more efficient than standard rTMS. In accordance with the approved treatment protocol, patients experience considerable sensory discomfort at a stimulation intensity of 120% of their resting motor threshold (rMT). Antidepressant effects of iTBS are believed to be mediated by modulating prefrontal excitability. There is still a lack of evidence to support the choice of 120% rMT as the optimal stimulation intensity, and the presumed superiority of higher stimulation intensities over lower intensities has yet to be proven. This knowledge gap has clinical implications since more tolerated treatments may lead to greater adherence, resulting in improved outcomes.

The current study proposes a randomized, triple-arm, controlled trial to compare the efficacy of iTBS at 75% (iTBS75) and 120% (iTBS120) rMT with sham iTBS (SiTBS). Based on the following considerations, SiTBS was selected to be compared with iTBS75 and iTBS120: SiTBS will reveal placebo antidepressant effects and serve as a control. iTBS75 is selected because iTBS at 80% aMT exhibits significant excitatory effects on the motor cortex and corresponds to approximately 70% rMT. There is however, a distance of about 12.7mm between the coil and the motor cortex, whereas 14.4mm separates the coil from the dorsolateral prefrontal cortex (DLPFC). Accordingly, a resting motor threshold of 70% at the motor cortex corresponds to a distance-adjusted rMT of 75% at the DLPFC. Lastly, iTBS120 is chosen as the standard stimulation intensity in current iTBS depression trials.

It is our intention to investigate the potential antidepressant effects of iTBS treatment at a much lower stimulation intensity than the one currently employed by most centers in the United States and approved in these centers. Thus, our study can contribute to establishing a treatment regimen with increased adherence and lower withdrawal rates.

DETAILED DESCRIPTION:
Introduction:

Key issues and knowledge gaps Intermittent theta-burst stimulation (iTBS), a special form of patterned repetitive transcranial magnetic stimulation (rTMS) approved by the U.S. Food and Drug Administration in 2018, is frequently used in many hospitals worldwide for the treatment of major depressive disorder (MDD). For example, at the Department of Psychiatry and Psychotherapy, Medical University of Vienna, the investigators perform about four iTBS treatments daily, amounting to about 1000 treatments a year. iTBS is safe, effective even in depressed patients that are refractory to standard pharmacological treatments, and has the advantage of increased efficiency over standard rTMS. The approved treatment protocol involves a stimulation intensity of 120% of the individual's resting motor threshold (rMT), an intensity associated with considerable sensory discomfort for patients.

The application of a stimulation intensity of 120% rMT is common practice in many psychiatric TMS clinics, and is based on research with conventional rTMS indicating higher clinical efficacy with higher stimulation intensity . However, neuroplastic effects of iTBS of the motor cortex are generally observed at much lower intensities. Researchers have observed significant excitatory effects of iTBS when the intensity is 80% of active motor threshold (aMT), which is approximately 70% of reactive motor threshold (rMT). Moreover, the assumption that the neuromodulatory effects are greater with increasing stimulation intensity is highly debated, and recent research indicates that a linear dose-response relationship for prefrontal iTBS is unfounded. Yet, modulation of prefrontal excitability is thought to underlie the antidepressant effect of iTBS. The investigators still lack evidence for the choice of 120% rMT as the optimal intensity and the presumed superiority of higher stimulation strengths over lower intensities is yet to be investigated. This is a knowledge gap that has important clinical implications because more tolerable treatments could result in greater adherence, and therefore ultimately better outcomes.

Here, the investigators propose a randomized, multicentre, triple-arm, controlled clinical trial to compare the efficacy of a 4-week treatment of daily iTBS at 75% (iTBS75) and 120% (iTBS120) rMT compared to sham iTBS (SiTBS). The choice to compare SiTBS with iTBS75 and iTBS120 is based on the following considerations: SiTBS will reveal placebo antidepressant effects and serves as a control condition. iTBS75 is chosen because iTBS at 80% aMT shows significant excitatory effects of the motor cortex and equals approximately 70% rMT. However, the distance from the coil to the motor cortex is on average 12.7mm whereas the distance to the dorsolateral prefrontal cortex (DLPFC) is about 14.4 mm. Hence, a resting motor threshold of 70% at the motor cortex corresponds to a distance-adjusted rMT of approximately 75% at the DLPFC. Finally, iTBS120 is chosen as it is the standard stimulation intensity in current iTBS trials for depression.

Our proposed study will elucidate the potential antidepressant effect of iTBS treatment at a much lower stimulation intensity than that currently employed by most centres and approved in the U.S. Hence, our study has a high potential to pave the way towards establishing a treatment regimen with increased adherence and lower rates of withdrawal.

Aims and Hypotheses to be tested:

This randomized, multicentre, triple-arm, controlled clinical trial aims to compare the efficacy of SiTBS with iTBS75 and iTBS120 after four weeks of daily treatments in patients with MDD. The investigators hypothesize that iTBS75 will be more effective in reducing depressive symptoms compared with SiTBS and iTBS120. More specifically, (1) the investigators hypothesize that the rate of response, defined as a reduction of Montgomery-Asberg Depression Rating Scale (MADRS) score to ≤50% of baseline values after treatment is significantly higher for iTBS75, compared to sham stimulation and iTBS120 (primary hypothesis). In a secondary analysis, the investigators will test the hypothesis that (2) the rate of remission, defined as a final MADRS score of ≤8, over the course of four weeks of treatment is significantly higher for iTBS75, compared to the other two arms. Similarly, the investigators hypothesise that the increase of (3) subjective mood and (4) happiness, assessed using PHQ-9 and SHS, respectively, is significantly higher for iTBS75, compared to the other two arms. Finally, the investigators hypothesize that (5) iTBS75 is more tolerable than iTBS120, as indicated by a lower reported pain sensation during iTBS75 compared to iTBS120.

ELIGIBILITY:
Inclusion Criteria:

* are aged between 18 and 70;
* have a MDD diagnosis, single or recurrent episode, diagnosed according to Diagnostic and Statistical Manual of Mental Disorders, fifth edition criteria and confirmed by means of the Mini-International Neuropsychiatric Interview (MINI);
* have a score of at least 18 on the 17-item Hamilton Rating Scale for Depression (HDRS17) in their current episode;
* have failed to have a clinically significant response to two or more standard antidepressant treatments during their current episode;
* have received stable psychopharmacological treatment within 4 weeks prior to screening; and
* have normal thyroid function, Complete Blood Count, electrolytes, and liver enzyme levels based on pre-study blood work.

Exclusion Criteria:

* have a history of substance abuse or dependence in the past 3 months;
* have a concomitant major unstable medical illness, cardiac pacemaker or implanted medication pump;
* show active suicidal intent (MADRS item 10 score >4);
* are pregnant;
* have a lifetime MINI diagnosis of bipolar I or II disorder, schizophrenia, schizoaffective disorder, schizophreniform disorder, delusional disorder, or current psychotic symptoms;
* have a metal implant or any other common MRI and TMS exclusion criteria;
* take antiepileptic drugs or benzodiazepines corresponding to a dose of >1 mg lorazepam per day;
* have had initiation or dose change of any psychotropic medication in the 4 weeks prior to screening or
* have undergone TMS in the past.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 246 (Estimated)
Dates: Start 2024-01-08 (Actual); Primary Completion 2026-04-26 (Estimated); Study Completion 2026-10-26 (Estimated)

PRIMARY OUTCOMES:
Montgomery-Asberg depression rating scale (MADRS) | through study completion, an average of 1 month
  The Montgomery-Åsberg Depression Rating Scale is a ten-item diagnostic questionnaire which psychiatrists use to measure the severity of depressive episodes in patients with mood disorders. Response rate after treatment (Montgomery-Asberg depression rating scale, MADRS reduction ≥50% of baseline)
  0 to 6: normal /symptom absent. 7 to 19: mild depression. 20 to 34: moderate depression. 35 to 60: severe depression.

SECONDARY OUTCOMES:
Patient Health Questionnaire-9 (PHQ-9) | through study completion, an average of 1 month
  The nine-item Patient Health Questionnaire is a depressive symptom scale
  PHQ-9 scores of 5, 10, 15, and 20 represented mild, moderate, moderately severe, and severe depression, respectively.
Subjective Happiness Scale (SHS) | through study completion, an average of 1 month
  The Subjective Happiness Scale seeks to conduct a global, subjective assessment of whether a person is happy or unhappy.
  A final score of subjective happiness is calculated by averaging the responses to the four items, with the 4th item's response being reverse coded (i.e., 7 turns to a 1, 6 turns to a 2, etc.). The final scores range from 1.0 to 7.0. Higher scores reflect greater subjective happiness.
Verbal Analogue Scale (VAS) Pain level | through study completion, an average of 1 month
  To ensure tolerability, the stimulation intensity will be adaptively titrated upward during the initial sessions of treatment to the target intensity without exceeding pain levels of 7, rated on a verbal analogue scale (VAS) ranging from 0 (no pain) to 10 (intolerable pain).

CONTACTS AND LOCATIONS:
Overall Officials: Georg Kranz, PhD, Principal Investigator — The Hong Kong Polytechnic University
Locations (1):
- The Hong Kong Polytechnic University, Hong Kong, Hong Kong

IPD SHARING:
Plan to Share IPD: No

DOCUMENTS (1):
  • Informed Consent Form (2024-01-01): https://cdn.clinicaltrials.gov/large-docs/67/NCT06392867/ICF_000.pdf